CLINICAL TRIAL: NCT00788788
Title: PoC Study of Heliox With Helium-Fractions Between 25 and 75% in Experimental Upper Airway Obstruction
Brief Title: Heliox in Experimental Upper Airway Obstruction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Dr. Hubert Trubel, University of Witten/Herdecke
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Heliox-PoC; EudraCT-No. 2006-005289-37
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-11

CONDITIONS: Airway Obstruction; Dyspnea
Keywords: Airway obstruction; Heliox; Different Helium content
MeSH Terms: conditions — Airway Obstruction; Dyspnea | interventions — heliox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Study subjects where breathing Heliox with a fraction of Helium of 25% followed by 50% and 75% with larger external resistor in comparison to medical air
  Interventions: Drug: HELIOX
- 2 (Active Comparator): Study subjects where breathing Heliox with a fraction of Helium of 50% followed by 75% and 25% with larger external resistor in comparison to medical air
  Interventions: Drug: HELIOX
- 3 (Active Comparator): Study subjects where breathing Heliox with a fraction of Helium of 25% followed by 50% and 75% with larger external resistor in comparison to medical air
  Interventions: Drug: HELIOX

INTERVENTIONS:
Drug: HELIOX — HELIOX is a mixture of Helium in Oxygen with a low density and the ability to reduce the work of breathing in subjects with airway obstruction. The fractions of Helium was altered in a different order depending on the arm of the study

SUMMARY:
Currently it is common medical wisdom that HELIOX (mixture of Helium in Oxygen) with a fraction of Helium below 60% is not effective in reducing airway obstruction. The investigators test the hypothesis that HELIOX with a fraction of Helium below 60% is still effective in relieving airway obstruction in a double-blind, randomized and controlled clinical PoC study with experimental upper airway obstruction.

DETAILED DESCRIPTION:
HELIOX is a mixture of Helium and Oxygen. It is a therapeutic modality that can improve upper and lower airway obstruction. The lower density of Helium can help to relieve airway obstruction and is known to lower the work of breathing. The fraction of Helium (FHe) in HELIOX should be maximized (e.g. up to a fraction of 79% with 21% of oxygen added) in order to achieve optimal anti-obstructive outcome and according to the literature a FHe below 60% renders HELIOX ineffective.

Objective: We conducted an investigator-initiated trial using different mixtures of Helium and Oxygen in 44 healthy volunteers in a randomized and double-blinded fashion.

Methods: After an adjustment phase the subjects were breathing through two different external resistors (intratracheal tube with inner diameter of either 4.0mm or 5.0mm) while gas of different composition (medical air with 79% Nitrogen and 21% Oxygen as control gas and HELIOX with a fraction of either 25%, 50% or 75% Helium in Oxygen, respectively) was provided in a blinded and random fashion. A crossover design was used so that every subject was exposed to every HELIOX gas mixture. Subjects were asked to score their degree of dyspnea after breathing different gas mixtures for 2 minutes intervals. In addition the variability of different hemodynamic parameters was assessed (continuous non-invasive blood pressure (systolic, diastolic and mean blood pressure), impedance cardiography (stroke volume and cardiac output), ECG (heart rate variability)) were assessed non-invasively and used to detected a change in the degree of airway obstruction in respect to the added load and the gas mixture.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes were recruited via posting in student forum of University of Witten/Herdecke
* Willingness to spend about 2h in the clinical exp. lab.

Exclusion Criteria:

* Acute airway infection
* History of asthma
* Smokers
* Pregnancy
* Abnormal lab. screen with liver function tests, Creat./BUN, CBC, blood glucose
* Anxiety or mood disorder
* Any chronic disease (incl. lung & heart disease, cancer, endocrine disorder)
* Mental retardation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Dyspnea score | Minutes
Variability of systolic blood pressure | Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Trubel, MD, Principal Investigator — University of Witten/Herdecke
Locations (1):
- HELIOS-Klinikum / University of Witten/Herdecke, Wuppertal, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Truebel H, Wuester S, Boehme P, Doll H, Schmiedl S, Szymanski J, Langer T, Ostermann T, Cysarz D, Thuermann P. A proof-of-concept trial of HELIOX with different fractions of helium in a human study modeling upper airway obstruction. Eur J Appl Physiol. 2019 May;119(5):1253-1260. doi: 10.1007/s00421-019-04116-7. Epub 2019 Mar 8. PMID 30850876